CLINICAL TRIAL: NCT04793477
Title: Comparison and Effectiveness of the Manual File System, the Multi-file Rotating System and the Single File Reciprocating System in Temporal Molars
Brief Title: Effectiveness of Rotating System and Single File Reciprocating System in Temporal Molars
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat Internacional de Catalunya (Other)
Responsible Party: Principal Investigator, Francisco Guinot-Jimeno, head of the department of pediatric dentistry, Universitat Internacional de Catalunya
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UIC-ODP-LIMAS
Record Dates: First submitted 2021-01-29; First posted 2021-03-11 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-04

CONDITIONS: Pulp Disease, Dental
Keywords: Pulpectomy; Rotary files; Reciprocating files
MeSH Terms: conditions — Dental Pulp Diseases | interventions — Pulpectomy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- K files (Dentsply Caulk, Milfors, DE, USA) (Experimental): Instrumentation with manual files shall be performed with balanced forces (Roane) technique consist of placing the instrument as apically as it can go and then turning it clockwise (less than 180º). This is followed by a counterclockwise rotation (of at least 120º) with slight apical pressure. This is repeated until the desired working length is obtained.
  Interventions: Device: instrumentation technique in pulpectomies
- VDW.ROTATE (VDW, Munich, Germany). (Experimental): Instrumentation with VDW.ROTATE files shall be performed with a glide path to WL using VDW.ROTATETM 15.04 until reaching working length (1.3cNm and 300-400 rpm), the next instrument in the sequence is VDW.ROTATETM 20.05 until reaching working length (2.1cNm and 300-400rpm). and finally instrument with VDW.ROTATETM 25.04 (2.3cNm and 300-400rpm)
  Interventions: Device: instrumentation technique in pulpectomies
- Reciproc® blue (RCP, VDW, Munich, Germany) (Experimental): Instrumentation with Reciproc blue files shall be performed with only one file and move it in a pecking motion (the amplitude will not exceed 3mm). All the instruments shall be cleaned after 3 pecks.
  Interventions: Device: instrumentation technique in pulpectomies

INTERVENTIONS:
Device: instrumentation technique in pulpectomies — comparison of three file systems for pulpectomies in primary molars

SUMMARY:
Is an in vivo study to test the effectiveness of the reciprocating system Reciproc blue and the rotating system VDW.ROTATE in primary molars.

DETAILED DESCRIPTION:
It is a randomized controlled clinical study to be conducted in the Department of Pediatric Dentistry of the International University of Catalonia (UIC).

The clinical study and data collection will be obtained by the second year students of the master's degree in Pediatric Dentistry. All of them will receive the same practical and theoretical training on the treatment to be performed, and will be calibrated by the principal investigator. The procedure and the data obtained will be reviewed by a trained investigator and blinded with the type of procedure used.

Children from 4 to 8 years old will be selected to visit the Clinica Universitaria de Odontología (CUO) with the master's degree in Pediatric Dentistry. A sample of 60 children will be taken. There will be three study groups, where 20 subjects will be assigned to each, estimating a follow-up loss ratio of 20%.

Once the patient is selected, they will be assigned to one of the groups in order of arrival. For example, patient one will be assigned in group 1, patient two in group 2, patient three in group 3 and so on.

There are 3 study groups groups: Group 1, with Manual instrumentation with K files (Dentsply Caulk, Milfors, DE, USA); group 2, with the VDW.ROTATETM (VDW, Munich, Germany); and group 3, with Reciproc® Blue (RCP, VDW, Munich, Germany) system.

A preliminary clinical and radiographic examination with periapical radiographs will be performed. To anesthetize the tooth, the student will use topical anesthesia (Urricaine gel, Clarben SA Laboratories) and local anesthesia with articaine 4% 1:200,000 epinephrine (Ultracaine; Normon S.A., Madrid, Spain) using a lower alveolar nerve block. The student will work with absolute isolation with rubber dam. The cavities will be removed with a high-speed diamond ball cutter and once the operator are inside the pulp chamber, will continue to remove the coronal pulp with a endo-Z cutter.

The operator will determine the working length (LT) with the Gold Reciproc motor (VDW, Munich, Germany), using K #15 file. LT is to be determined it at 1 mm less than what the locator indicates due to the physiological reabsorptions present in the tooth. Each group will be instrumented according to the manufacturer's instructions, explained above. The duct permeability will be ensured with K #10 file with between files and at the end of the instrumentation. The duct irrigation was carried out with 5ml of 2,5% NaOCl in each duct and a side outlet needle. In the case of group 3, which is a single lime system, the operator will take into account that the irrigation must be similar to that of the other systems.

Once the instrumentation is finished,the elapsed time will be recorded from the beginning to the end of the instrumentation with the disinfection of the appropriate irrigant. The operator will record the minutes and seconds evaluated with an analog stopwatch. The ducts will be dried with sterile paper tips and place the sealing material, calcium hydroxide with iodophormic paste (Vitapex; Neo Dental International Inc., Federal Way, WA, USA). The sealing material will be placed with the applicator tip that comes with the product and at the end we will compact the sealing with a cotton ball in the chamber. The application material procedure will be carried out in this way, to know if the success of the sealing depends on the system of files used. The tooth will remain with a temporary Eugenol Zinc Oxide (IRM; Dentsply Caulk, Milfors, DE, USA) filler until the next visit, which will be a week later, to place a stainless steel crown (3M ESPE, St. Paul, MN, USA) cemented with glass ionomer cement (Ktac-Cem;3M ESPE, St. Paul, MN, USA).

To finish the treatment, a periapical radiography will be done to the patient. With the final periapical radiography, a researcher blinded to the study groups, will evaluate the quality and quantity of the seal without the need for auxiliary elements such as léntulos or files. The filling will be evaluated if it's optimal, under-filled, over-filled or with the presence of gaps.

To determine the patient's anxiety during dental treatment, the operator will use a pulse oximeter (digital Onyx, NONIN, Plymouth, MN, USA). The child's heart rate will be evaluated in the following moments: 3 min before the application of topical anesthesia, at the topical anesthesia aplication, during the application of the local anesthetic, when the rubber dam is placed, during the instrumentation and removal of coronal pulp tissue, during the instrumentation with each file system, and finally when the rubber dam is removed. The average heart rate will be determined for each period by a set of values in a period of 1 minute.

At the end of the treatment the operator will evaluate the behavior of the child with the Frankl scale where 1 is very uncooperative and 4 is very collaborative; and will see if it is similar to the behavior of previous visits with conservative treatment.

To determine the ease of operation, a numerical scale from 0 to 10 is will be used, where 0 means very easy to use and 10 very difficult. It will be taken into account that if there are more than one operator, they have the same acquired skills and the same familiarity with the file systems used.

In the evaluation of postoperative pain, that same day the patient's parents will be given a questionnaire where the parents will have to write down at 6, 12, 24, 48, 72 hours and a week later, the pain felt. The pain will be evaluated with the Wong-Baker scale because facial scales are usually easier for the pediatric patient. All patients will be given a 2% junifen prescription with a weight-appropriate dose in case of postoperative pain. Parents will be advised that the prescription should only be used in cases of more severe pain, and will need to be noted on the data collection sheet. When these patients need taking medication, the marked value at the Wong-Baker station will not be taken into account. It will be noted that they are patients who have required medication. The operator will collect the data a week, coinciding with the stainless steel crown placement.

All the data obtained from the patients participating in the study will be recorded in two sheets: One for the operator, where the age, sex, the assigned study group, and all the variables studied will be recorded: instrumentation time, filler quality, operator's ease, behavior and anxiety of the patient; The other sheet will be for parents to record at home the postoperative pain felt by the child.

Statistical analysis will be caried out with Statgraphics Plus 5.1 version and Microsoft Excel.

An absolute and relative frequency shall be used in categorical variables to describe the data. For the numerical variables the mean and standard deviation or median and first and third quartile will be used, depending on whether the data is parametric or not. To be able to make comparisons between files, the Chi-square T will be used for categorical variables and the T-student or Mann Whitney test for numerical variables. The SHAPIRO WILKS contrast will be used to compare the normality of the data.

For this study, a 95% confidence interval is to be taken into account, taking as statistically significant reference a p value ≤ 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Vital or non-vital temporary lower second molars.
* Radiographic absence of external or internal pathological reabsorption.
* Absence of interadicular radioluscience and/or periapical lesion.
* Temporary teeth with at least 2/3 of the root intact or a minimum root length of 8mm.
* Remaining dental structure sufficient for the subsequent placement of a stainless steel crown.
* Children who have already undergone some previous restorative treatment in the Department of Pediatric Dentistry.

Exclusion Criteria:

* Molars that have less than 2/3 radicular lenght.
* Have taken analgesics or anti-inflammatories in the last 12 hours.
* Very uncooperative patients, who require some type of anxiety to be treated.
* Patients with systemic diseases.
* Patients with special needs.

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Evaluate instrumentation time with K, Rotate and Reciproc Blue files. | Immediately after instrumentation. From the beginning to the end of the instrumentation with the files
  Once the instrumentation and irrigation is finished, the operator will record the time elapsed from the beginning to the end of the instrumentation with the disinfection of the appropriate irrigant. The operator will record the minutes and seconds evaluated with an analog stopwatch.

SECONDARY OUTCOMES:
Evaluate the postoperative pain with the K files, the Rotate and the Reciproc Blue. | at 6, 12, 24, 48, 72 hours and a week later
  In the evaluation of postoperative pain, that same day the patient's parents will be given a questionnaire where they will have to write down at 6, 12, 24, 48, 72 hours and a week later, the pain felt. The pain will be evaluated with the Wong-Baker scale because facial scales are usually easier for the pediatric patient.The scale goes from 0 to 10, where 0 means no pain and 10 means the worst possible pain. All patients will be given a 2% junifen prescription with a weight-appropriate dose in case of postoperative pain. Parents will be advised that the prescription should only be used in cases of more severe pain, and will need to be noted on the data collection sheet. When these patients need taking medication, the marked value at the Wong-Baker station will not be taken into account. It will be noted that they are patients who have required medication.
Evaluate the quality of the filling of the duct without the need of any auxiliary elements with the files K, the Rotate and the Reciproc Blue. | Immediately after the procedure
  A periapical radiography will be done to the patient. With the final periapical radiography, a researcher blinded to the study groups, will evaluate the quality of the seal without the need for auxiliary elements. The filling will be evaluated if it's optimal, under-filled, over-filled or with the presence of gaps.
Evaluate the child's behavior comparing to some previous restorative treatment with K, Rotate and Reciproc Blue files. | Immediately after the procedure
  At the end of the treatment the operator will evaluate the behavior of the child with the Frankl scale where 1 is very uncooperative and 4 is very collaborative; and the operator will see if it is similar to the behavior of previous visits with conservative treatment.
Evaluate the child's heart rate during instrumentation with K, Rotate and Reciproc Blue files. | During one week. Evaluation 3 minutes before topical anesthesia, topical anesthesia, local anesthesia, rubber dam, caries removal and coronal pulp tissue elimination, duct instrumentation, rubber dam removed.
  The operator will use a pulse oximeter (digital Onyx, NONIN, Plymouth, MN, USA). The child's heart rate will be evaluated in the following moments: 3 minutes before the application of topical anesthesia, at the topical anesthesia aplication, during the application of the local anesthetic, when the rubber dam is placed, during the instrumentation and removal of coronal pulp tissue, during the instrumentation with each file system, and finally when the rubber dam is removed. The average heart rate will be determined for each period by a set of values in a period of 1 minute.
Evaluate the operator ease during instrumentation with K, Rotate and Reciproc Blue files. | Immediately after the procedure
  To determine the ease of operation, the researcher use a numerical scale from 0 to 10, where 0 means very easy to use and 10 very difficult. It will be taken into account that if there are more than one operator, they have the same acquired skills and the same familiarity with the file systems used

CONTACTS AND LOCATIONS:
Locations (1):
- Universitat Internacional de Catalunya, Sant Cugat del Vallès, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No